CLINICAL TRIAL: NCT03389347
Title: Individualized Treatment for Relapsed/Refractory Multiple Myeloma Based on High Throughput Drug Sensitivity and Genomics Data
Brief Title: High Throughput Drug Sensitivity and Genomics Data in Developing Individualized Treatment in Patients With Relapsed or Refractory Multiple Myeloma or Plasma Cell Leukemia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9944; NCI-2017-02204 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9944 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1017011 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-12-11; First posted 2018-01-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-02

CONDITIONS: Plasma Cell Leukemia; Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Leukemia, Plasma Cell; Multiple Myeloma | interventions — High-Throughput Screening Assays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device feasibility (high-throughput assay, sequencing) (Experimental): Patients undergo collection of bone marrow aspirate and blood for high-throughput drug sensitivity assay and mutational analysis using next generation sequencing. Patients and their treating physicians receive the results of the tests. Treatment decisions are then made by the patients and their treating physicians.
  Interventions: Procedure: Biospecimen Collection; Device: High Throughput Screening; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of bone marrow aspirate and blood
Device: High Throughput Screening — Anti-tumor drugs are tested against myeloma cells in the laboratory, in a high-throughput drug sensitivity assay
  Other Names: High Throughput Assay
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies whether using high throughput drug sensitivity and genomics data is feasible in developing individualized treatment in patients with multiple myeloma or plasma cell leukemia that has come back or does not respond to treatment. High throughput screen tests many different drugs that kill multiple myeloma cells in individual chambers at the same time. Matching a drug or drug combination to a patient using high throughput screen and genetic information may improve the ability to help patients by choosing drugs that work well for their disease.

DETAILED DESCRIPTION:
OUTLINE:

Patients undergo collection of bone marrow aspirate and blood for high-throughput drug sensitivity assay and mutational analysis using next generation sequencing. Patients and their treating physicians receive the results of the tests. Treatment decisions are then made by the patients and their treating physicians.

After completion of study, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma or plasma cell leukemia with documented relapsed or refractory disease according to International Myeloma Working Group (IMWG) criteria, in any one of the following categories:

  * 3 prior lines of therapy including an immunomodulatory drug (IMiD) and a proteasome inhibitor (PI)
  * Less than a very good partial response (VGPR) to initial therapy
  * Early relapse (< 12 months) after autologous hematopoietic cell transplant (HCT) or after 1st line of therapy
* Collection of a bone marrow, fluid or tissue sample that is expected to have enough cells to run the assay
* Measurable disease defined by one of the following:

  * Serum monoclonal protein >= 0.5 g/dL by serum protein electrophoresis (SPEP)
  * >= 200 mg/monoclonal protein in urine on 24 hr urine protein electrophoresis (UPEP)
  * Involved serum free light chain (FLC) >= 10 mg/dL and abnormal involved:uninvolved ratio
  * Plasma cytomas that are palpable per exam or measurable per standard radiologic review
  * Circulating plasma cells >= 2,000 if diagnosis of plasma cell leukemia
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-3
* Female patients of child bearing potential and non-vasectomized male patients agree to practice appropriate methods of birth control
* Ability to understand purpose and risks of the study and provide signed and dated informed consent, and authorization to use protected health information
* Expected survival is > 100 days
* Adequate organ function as determined by the investigator

Exclusion Criteria:

* Mucosal or internal bleeding, or platelet transfusion refractory
* Any medical conditions that would impose excessive risk to the patient, or would adversely affect his/her participation in the study
* Known active infection requiring antibiotics within 7 days of initiation of study treatment, unless considered controlled in the opinion of the investigator
* Other malignancy with life expectancy < 1 year due to the other malignancy
* Pregnant or breast feeding women
* Serious psychiatric illness, alcoholism, or drug addiction
* Human immunodeficiency virus (HIV), or active hepatitis B or C infection
* Previous treatments for multiple myeloma (MM) within 2 weeks of initiation of study treatment
* Prior autologous or allogeneic stem cell transplantation (SCT) within 12 weeks of initiation of study treatment
* Prior allogeneic hematopoietic cell transplantation (HCT) with active graft versus host disease (GVHD) on therapeutic dosing of immunosuppression or prednisone > 20 mg daily equivalent
* Prior major surgical procedure or radiation treatment within 2 weeks of initiation of study treatment (not including limited radiation used for palliation of bone pain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Actionable assay result | Up to 21 days
  The feasibility of this approach will be assessed in terms of obtaining an actionable response from the proposed assay in at least 50% of patients examined.

SECONDARY OUTCOMES:
Overall response rate to the therapy chosen after performing the assay | Up to 2 years
  Will be assessed by the International Myeloma Working Group (IMWG) response criteria. The response among all patients who received the assay as well as among patients who obtained an actionable result from the assay will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Danai Dima, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No